CLINICAL TRIAL: NCT02153294
Title: PRotective VENTilation in Patients Without ARDS at Start of Ventilation - PReVENT, a Randomized Controlled Trial
Brief Title: PRotective VENTilation in Patients Without ARDS
Acronym: PReVENT-NL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Tergooi Hospital (Other); Leiden University Medical Center (Other); Gelre Hospitals (Other); Amsterdam UMC, location VUmc (Other); Westfries Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Principal Investigator and Clinical Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PReVENT-NL; 80-83700-98-42001 (Other Grant/Funding Number: 2013/16475/ZONMW)
Record Dates: First submitted 2014-05-23; First posted 2014-06-03 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Ventilator-free Days
Keywords: low tidal volume; high tidal volume; protective ventilation; ARDS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ventilation with lower tidal volumes (Experimental): Use of low tidal volume (4 to 6 ml/kg PBW) after intubation and during all mechanical ventilation
  Interventions: Procedure: low tidal volume
- Ventilation with higher tidal volumes (Other): Use of high tidal volume (8 to 10 ml/kg PBW) after intubation and during all mechanical ventilation
  Interventions: Procedure: high tidal volume

INTERVENTIONS:
Procedure: low tidal volume — Patients are randomized and ventilated with a low tidal volume (4-6 ml/kg PBW)
  Arms: Ventilation with lower tidal volumes
Procedure: high tidal volume — Patients are randomized and ventilated with a high tidal volume (8-10 ml/kg PBW)
  Arms: Ventilation with higher tidal volumes

SUMMARY:
The purpose of this national multicentre randomized controlled trial is to compare a ventilation strategy using lower tidal volumes and higher respiratory rates with a ventilation strategy using higher tidal volumes and a lower respiratory rate in intubated and ventilated intensive care unit (ICU) patients without Acute Respiratory Distress Syndrome (ARDS) at start of ventilation.

Participating centres in The Netherlands will include a total of 952 adult patients admitted to intensive care units without ARDS. Patients are randomized and ventilated with either a strategy with lower tidal volumes (4 to 6 ml/kg predicted body weight (PBW)) or a strategy with higher tidal volumes (8 to 10 ml/kg PBW). Patients will be assessed every day until day 28 or discharge of the intensive care unit, whichever comes first, on day 28 and on day 90. Primary endpoint is the number of ventilator-free days at day 28. Secondary endpoints are ICU- and hospital length of stay (LOS) and - mortality, the incidence of development of ARDS, pneumonia, atelectasis, and pneumothorax, the cumulative use and duration of sedatives, and neuromuscular blocking agents, incidences of ICU delirium and ICU acquired weakness, patient-ventilator asynchrony and the need for decreasing of instrumental dead space.

DETAILED DESCRIPTION:
Research question:

Does mechanical ventilation with lower tidal volumes, as compared with mechanical ventilation with higher tidal volumes, increase the number of ventilator-free days at day 28 in patients without ARDS at start of ventilation?

Study Design:

An investigator-initiated, national, multicenter, parallel randomized controlled two-arm trial.

Centers:

Five centers in The Netherlands will participate in this trial;

* Academic Medical Center, University of Amsterdam
* Gelre Hospitals, Apeldoorn
* Leiden University Medical Center, Leiden
* Tergooi, Hilversum
* Vrije Universiteit University Medical Center, Amsterdam
* Westfries Gasthuis, Hoorn

Ethics Approval: The Institutional Review Board of the Academic Medical Center approved of the study on 15 May 2014

Monitoring:

* Monitoring of patients safety and reviewing of safety issues is performed by a designated independent Data Safety and Monitoring Board (DSMB).The DSMB watches over the ethics of conducting the study in accordance with the Declaration of Helsinki. This study compares two treatment strategies that are used in standard care, therefore no related serious adverse events (SAEs) are expected. All unexpected and related or possibly related adverse events will be reported to the DSMB
* An independent monitor will perform clinical trial monitoring. On-site monitoring will comprise controlling presence and completeness of the research dossier and the informed consent forms, source data checks will be performed. Every participating center will be visited at least once every year.

Study Population:

Adult ICU-patients without ARDS with an expected duration of ventilation longer than 24 hours, within 1 hour after initiation of ventilation or admittance to the ICU if already intubated and ventilated on admission.

Sample Size Calculation:

The required sample size is calculated using data from the recently published meta-analysis and a secondary analysis of this meta-analysis using individual patient data from the studies performed in ICU patients [submitted for publication]. The sample size is computed on the basis of the hypothesis that ventilation with lower tidal volumes is associated with a reduction of one day of ventilation. A sample size of 397 patients in each group has 80% statistical power to detect a difference of one ventilator-free day and alive at day 28 after ICU admission, with means of 23 and 24 days respectively. Assuming that the common standard deviation is 5 using a two group t-test with a 0.05 two-sided significance level. The sample size is increased by 20% to correct for dropouts and lost to follow up (i.e., because patients could be transferred to other hospitals), meaning that each group will contain 476 patients.

Methods:

Patients in participating intensive care units (ICU) are screened and randomized within 1 hour of start of mechanical ventilation in the unit. Demographic data on screened patients regardless of meeting enrollment criteria will be recorded (registry: age, gender, type of surgery). Randomization will be performed using a dedicated, password protected, SSL-encrypted website. Randomization sequence is generated by a dedicated computer randomization software program using random block sizes and is stratified per center and per intubation location (i.e., in the ICU or before ICU admittance in the operation room or in the emergency room). No blocking is applied to other trial factors. Due to the nature of the intervention, blinding is not possible.

Patients are randomly assigned in a 1:1 ratio to lower tidal volume ventilation (4 to 6 ml/kg PBW) (the 'lower tidal volume'-arm) or ventilation with higher tidal volumes (8 to 10 ml/kg PBW) (the 'higher tidal volume'-arm).

The allowed ventilation modes are volume controlled ventilation and pressure support ventilation. The inspiration-to-expiration ratio with volume controlled ventilation is 1:2. With volume controlled ventilation the inspiration time and pause are set at 25% and 10% respectively. With pressure support ventilation the highest possible pressure rise is chosen, and cycling off is set at 25%. The inspired oxygen fraction is 0.21 or higher to maintain oxygen saturation 90 to 92% and/or PaO2 > 7.3 to 10.7 kPa (55 to 80 mmHg). The respiratory rate is adjusted to maintain a blood pH of 7.25 to 7.45. In case of metabolic acidosis or - alkalosis, a lower or higher than normal PaCO2 can be accepted, left to the discretion of the attending physician. The lowest level of positive end-expiratory pressure is 5 cmH2O. Recruitment maneuvers are allowed, when deemed necessary, left to the discretion of the attending physician. In both arms a tidal volume is titrated per PBW, which is calculated according to a previously used formula: 50 + 0.91 x (centimeters of height - 152.4) for males and 45.5 + 0.91 x (centimeters of height - 152.4) for females.

* Patients randomized to the 'lower tidal volume'-arm start with a tidal volume of 6 ml/kg PBW. The tidal volume size is decreased in steps of 1 ml/kg PBW per hour, to a minimum of 4 ml/kg PBW, unless the patient suffers from severe dyspnea (identified by increased respiratory rate > 35 breaths per minute accompanied by increasing levels of discomfort with or without need for more sedation) or unacceptable acidosis.The following measures can be taken to prevent respiratory acidosis: increasing respiratory rate and decreasing instrumental dead space by shortening ventilation tubing, to limit dead space ventilation. Patients randomized to the lower tidal volume arm may need very little support when the ventilator is switched to pressure support ventilation, but a minimum of 5 cmH2O should be used. In case the resulting tidal volume exceeds 6 ml/kg PBW this must be accepted
* Patients randomized to the 'higher tidal volume'-arm start with a tidal volume of 10 ml/kg PBW. With volume-controlled ventilation the plateau pressure should not exceed 25 cm H2O. Only if the plateau pressure exceeds 25 cm H2O the tidal volume is decreased in steps of 1 ml/kg PBW per hour, to a minimum of 8 ml/kg PBW (table 1). With pressure support, tidal volume titration is by variation of the pressure support level. Other modes of ventilation are not allowed.Patients randomized to the higher tidal volume arm generally need more support when the ventilator is switched to pressure support ventilation, but the maximal airway pressure should not exceed 25 cm H2O [2]. In case the resulting tidal volume remains below 10 ml/kg PBW this must be accepted.
* Daily assessment of the ability to breathe with pressure support ventilation is required as soon as FiO2 ≤ 0.4 or when the PEEP level and FiO2 level are lower than the day before. Other modes of ventilation are not allowed.In addition, the ventilator can be switched to pressure support ventilation at any moment the attending nurse or physician consider the patient is awake enough to breathe with pressure support ventilation. Assessment of the ability to breathe with pressure support is also required in case patient-ventilator asynchrony is noticed (ineffective breathing; double triggering, use of assessory respiratory muscles). A patient is assumed to be ready for extubation when the following criteria are met for at least 30 minutes, the final decision for extubation is made by the attending physician:

  * Responsive and cooperative
  * Adequate cough reflex
  * PaO2/FiO2 of > 200 mmHg with FiO2 ≤ 40%
  * Respiratory rate of 8 to 30/minute
  * No signs of respiratory distress (i.e., marked accessory muscle use, abdominal paradox, diaphoresis, marked dyspnea)
  * Pressure support level < 7 cm H2O (lower tidal volume arm) or < 12 cm H2O (higher tidal volume arm)
  * Hemodynamically stable (systolic blood pressure 80 to 160 mmHg and heart rate 40 to 130/min) and no uncontrolled arrhythmia
  * Temperature > 36.0oC and < 38.5oC In the higher tidal volume arm physicians and nurses may decide to lower the pressure support level first (i.e., before extubation). For this, the pressure support level is lowered step-wise with steps of 2 to 5 cm H2O per hour to < 7 cm H2O. If this is not tolerated according to the conditions mentioned above, the pressure support level is set back to maintain a tidal volume as per randomization and the patient is assessed for extubation the following day. If a patient becomes able to breathe without assistance but subsequently requires additional ventilation within 28 days after randomization, the same tidal volume protocol is resumed. Non-invasive ventilation is allowed, but it should be tried to have comparable tidal volumes as with invasive ventilation, as per randomization.

Sedation follows the local guidelines for sedation in each participating units. In general, these guidelines favor the use of analgo-sedation over hypno-sedation, use of bolus over continuous infusion of sedating agents, and the use of sedation scores. Nurses determine the level of sedation at least 3 times per day. The adequacy of sedation in each patient is evaluated using a Richmond Agitation Sedation Scale (RASS). A RASS score of -2 to 0 is seen as adequate sedation. As stated above, sedation adjustments should never be done to allow a lower or higher tidal volume. The goals of sedation are to reduce agitation, stress and fear; to reduce oxygen consumption (heart rate, blood pressure and minute volume are measured continuously); and to reduce physical resistance to- and fear of daily care and medical examination. Patient comfort is the primary goal.

Statistical Analysis:

* The primary outcome, the number of ventilator-free days at day 28 after ICU admission, is analyzed using Cox's regression. Possible imbalance between groups will be modeled in the Cox model. P-values of 0.05 are used for statistical significance. When appropriate, statistical uncertainty will be expressed by the 95% confidence levels.
* Continuous normally distributed variables will be expressed by their mean and standard deviation or when not normally distributed as medians and their interquartile ranges. Categorical variables will be expressed as n (%). To test groups Student's t test will be used, if continuous data is not normally distributed the Mann-Whitney U test will be used. Categorical variables will be compared with the Chi-square test or Fisher's exact tests. Time dependent data will be analyzed using a proportional hazard model adjusted for possible imbalances of patients' baseline characteristics. Patient characteristics will be compared and described by appropriate statistics.
* The goal of the primary analysis is to quantify the effect of lower tidal volumes vs. higher tidal volumes on the number of ventilator free days and alive at day 28. Statistical analysis will be based on the intention-to-treat principle. We will also perform a per-protocol analysis, comparing patients who received lower tidal volumes and patients who received higher tidal volumes. Other secondary analyses include analysis of patients who had pneumonia versus patients without pneumonia, patients who fulfilled the definition for mild ARDS versus patients who did not fulfill this definition, and patients with sepsis versus patients without sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Admission to an ICU participating in this trial
* Need for intubation
* Within 1 hour of admission from the operation room or emergency room (if still intubated and ventilated), or within 1 hour of start of invasive ventilation in the ICU
* An expected duration of ventilation > 24 hours

Exclusion Criteria:

* Age less than 18 years
* Patients previously randomized in PReVENT
* Patients participating in other interventional trials
* Patients with a clinical diagnosis of ARDS according to the Berlin definition
* Patients with a PaO2/FiO2 < 200 mm Hg in whom hypoxia is presumably not caused by cardiac failure or fluid overload
* Invasive ventilation longer than 12 hours directly preceding admission
* Patients with suspected or confirmed pregnancy
* Patients with increased and uncontrollable intracranial pressure (of ≥18 mmHg)
* Patients with GOLD classification III or IV chronic obstructive pulmonary disease (COPD)
* Patients with asthmatic status
* Patients with premorbid restrictive pulmonary disease (evidence of chronic interstitial infiltration on previous chest radiographs)
* Patients with new proven pulmonary thrombo-embolism
* Patients with any previous pneumectomy or lobectomy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 952 (Actual)
Dates: Start 2014-08; Primary Completion 2017-09-20 (Actual); Study Completion 2017-11-18 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days | first 28 days after start of ventilation
  The number of ventilator-free days, defined as the number of days from day 1 to day 28 on which a patient breathes without assistance, if the period of unassisted breathing lasted at least 24 consecutive hours.

SECONDARY OUTCOMES:
Intensive care unit length of stay | first 90 days after start of ventilation
Hospital length of stay | first 90 days after start of ventilation
Cumulative use and duration of sedatives and neuromuscular blocking agents | first 28 days after start of ventilation or discharge from intensive care
ICU delirium | first 28 days after start of ventilation or discharge from intensive care
  Development of delirium according to the Confusion Assessment Method for intensive care unit (CAM-ICU)
ICU- Acquired Weakness | first 28 days after start of ventilation or discharge from intensive care
  Development of ICU-acquired weakness using the Medical Research Council (MRC) score and grip strength assessment
Mortality | first 90 days after start of ventilation
  Any death during ICU-, or hospital-stay and within 90 days
Pulmonary complications | first 28 days after start of ventilation or discharge from intensive care
  Development of ARDS according to the Berlin definition, pulmonary infection, atelectases and pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J Schultz, MD, PhD, Principal Investigator — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Fabienne D Simonis, MD, Study Director — Academic Medical Center, University of Amsterdam, The Netherlands; Marcelo Gama de Abreu, MD, PhD, Study Chair — Department of Anesthesiology and Intensive Care Medicine, University Hospital Carl Gustav Carus, Technical University Dresden, Germany; Paolo Pelosi, MD, PhD, Study Chair — Department of Surgical Sciences and Integrated Diagnostics, University of Genoa, Italy; Ary Serpa Neto, MD, MSc, Study Chair — Department of Intensive Care, Academic Medical Center, University of Amsterdam, The Netherlands; Janneke Horn, MD, PhD, Principal Investigator — Department of Intensive Care, Academic Medical Center, University of Amsterdam, The Netherlands; Nicole P Juffermans, MD, PhD, Principal Investigator — Department of Intensive Care, Academic Medical Center, University of Amsterdam, The Netherlands; Jan M Binnekade, PhD, Principal Investigator — Department of Intensive Care, Academic Medical Center, University of Amsterdam, The Netherlands; Gerard Innemee, MD, Principal Investigator — Tergooi, Hilversum, The Netherlands; Evert de Jonge, MD, PhD, Principal Investigator — Leiden University Medical Center, Leiden, The Netherlands; Peter E Spronk, MD, PhD, Principal Investigator — Gelre Hospitals, Apeldoorn, The Netherlands; Pieter Roel Tuinman, MD, PhD, Principal Investigator — VU Medical Center, Amsterdam, The Netherlands
Locations (1):
- Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam, Netherlands

REFERENCES:
- [Derived] van Meenen DMP, Algera AG, Schuijt MTU, Simonis FD, van der Hoeven SM, Neto AS, Abreu MG, Pelosi P, Paulus F, Schultz MJ; for the NEBULAE; PReVENT; RELAx investigators. Effect of mechanical power on mortality in invasively ventilated ICU patients without the acute respiratory distress syndrome: An analysis of three randomised clinical trials. Eur J Anaesthesiol. 2023 Jan 1;40(1):21-28. doi: 10.1097/EJA.0000000000001778. Epub 2022 Nov 18. PMID 36398740
- [Derived] Writing Group for the PReVENT Investigators; Simonis FD, Serpa Neto A, Binnekade JM, Braber A, Bruin KCM, Determann RM, Goekoop GJ, Heidt J, Horn J, Innemee G, de Jonge E, Juffermans NP, Spronk PE, Steuten LM, Tuinman PR, de Wilde RBP, Vriends M, Gama de Abreu M, Pelosi P, Schultz MJ. Effect of a Low vs Intermediate Tidal Volume Strategy on Ventilator-Free Days in Intensive Care Unit Patients Without ARDS: A Randomized Clinical Trial. JAMA. 2018 Nov 13;320(18):1872-1880. doi: 10.1001/jama.2018.14280. PMID 30357256
- [Derived] Simonis FD, Binnekade JM, Braber A, Gelissen HP, Heidt J, Horn J, Innemee G, de Jonge E, Juffermans NP, Spronk PE, Steuten LM, Tuinman PR, Vriends M, de Vreede G, de Wilde RB, Serpa Neto A, Gama de Abreu M, Pelosi P, Schultz MJ. PReVENT--protective ventilation in patients without ARDS at start of ventilation: study protocol for a randomized controlled trial. Trials. 2015 May 24;16:226. doi: 10.1186/s13063-015-0759-1. PMID 26003545